CLINICAL TRIAL: NCT05592834
Title: Effect of the Positive Deviance and Parent Facilitator Training Strategies to Malnutrition and Caregiving Among Children and Youth With CP in the Iganga, Mayuge and Bugweri Rural Districts of Eastern Uganda"
Brief Title: Caregiver Led Strategies to Malnutrition and Care-giving Among Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Makerere University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: HDREC 186
Record Dates: First submitted 2022-10-20; First posted 2022-10-25 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Weight Gain
MeSH Terms: conditions — Weight Gain

STUDY DESIGN:
Intervention Model Description: This will be a 2x2 factorial quasi-randomised controlled trial assessing the effects of the Positive deviance (PD) (Yes/No) and Parent facilitator training (PFT) (Yes/No) strategies within four experimental conditions: i) Both PD and PFT, ii) Only PD, iii)Only PFT, iv) Neither PD and nor PFT(controls).
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Evaluators, Participants, and caregivers facilitating the PFT and PD training sessions will be blinded on group allocations. A group of independent outcome assessors (evaluators), not involved in the intervention, will administer the outcome measures after the interventions. These evaluators will also be blinded to group allocation to avoid reporting bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Positive deviance (PD) (Experimental): This group will receive only the positive deviance intervention and not the PFT
  Interventions: Behavioral: positive deviance hearth strategy
- Parent facilitator training (PFT) (Experimental): This group will receive only the parent facilitator training intervention and not the PD
  Interventions: Behavioral: Parent facilitator trainings
- Parent facilitator and positive deviance(PFT/PD) (Experimental): This group will receive both the PD and PFT interventions
  Interventions: Behavioral: positive deviance hearth strategy; Behavioral: Parent facilitator trainings
- Control (Active Comparator): This group will receive neither the PD nor the PFT interventions but care as usual.
  Interventions: Other: Control

INTERVENTIONS:
Behavioral: positive deviance hearth strategy — The PD-program is run for 3-months with 2 weeks (12 days) of nutrition education and rehabilitation sessions (NERS) conducted in each month. Each day session includes an half hour education session and a one and half hour peer led cooking session. Caretakers learn how to rehabilitate their malnourished children under the supervision and the support of caregivers who have well-nourished children (positive deviants). Children are nutritionally assessed by trained nutrition assistants or clinician on the 1st day of the NERS sessions and after three months.
  During the rehabilitation sessions, caregivers learn how to prepare nutrient-rich meals for their children from locally available food identified during the positive deviance-inquiry, and actively practice good feeding and hygiene practices. Caregivers together prepare food menus based on the PD-inquiry good foods or what they can conveniently access but of equal nutritional value.
  Arms: Parent facilitator and positive deviance(PFT/PD); Positive deviance (PD)
Behavioral: Parent facilitator trainings — Primary caregivers of children with CP residing in the study setting are trained as parent facilitators by expert physical rehabilitation therapist . Trained parent facilitators then hold fellow caregiver workshops each lasting approximately two hours long and includes between 6-10 caregivers. To ensure quality and consistency of the workshops, the Parent Facilitators follow a detailed manual adapted from the Carer-2-Carer Programme translated into Lusoga, the local language. No expert therapists is involved in the parent facilitator training workshops. Parent facilitator training workshops involve 7 sessions that expose caregivers to understanding CP and how to improve body functioning: session1: what is CP? session2: CP as a way of life, Session 3: Getting my child's body ready to move, Session 4: Eating and drinking a healthy diet, Session 5: communication, Session 6: Play, and Session 7: Central visual impairment.
  Arms: Parent facilitator and positive deviance(PFT/PD); Parent facilitator training (PFT)
Other: Control — This group will receive neither the PD nor the PFT interventions but care as usual
  Arms: Control

SUMMARY:
The goal of this factorial trial is to test and compare the effectiveness of two caregiver led strategies, i.e., the positive deviance nutrition(PD) strategy and the parent facilitator training (PFT) strategies, to malnutrition and care-giving among children and youth with cerebral palsy. Participants will be assigned to receive either of the four conditions, including,

* PFT only,
* PD only,
* Both the PFT and PD,
* None of the PD or PFT (controls) Researchers will compare either groups to see if there is an improvement in the nutritional status by weight gain and care giving knowledge and practices

DETAILED DESCRIPTION:
High malnutrition and related mortality risk is common among children with cerebral palsy (CP) in most low- and middle-income countries. This is partly due to limited access to mainstream health care services worsened by the scarcity of health professionals with an extra skill in special needs care, including the ability to manage feeding difficulties common in the CP population. Families of children with CP have thus been left alone to care for their child without a clear direction on how to provide the best care including effective feeding and nutrition practices. This amplifies the relevance of caregivers in the improvement of CP child survival, and justifies the need for affordable and culturally acceptable strategies.

Training of caregivers of children with CP as lay professionals has become a cost-effective strategy to address the physical rehabilitation workforce gap in some African countries. However, the effectiveness of these strategies is not properly evaluated with regards to managing malnutrition in CP. Furthermore, caregiver-initiated strategies like the positive deviance nutrition strategy although proven effective in the management of malnutrition among typically developed children, its effectiveness in the CP child population is not clear. This study seeks to evaluate the effectiveness of caregiver led strategies i.e., the positive deviance and parent facilitator training (physical rehabilitation) strategies, to malnutrition and care-giving among children and youth with CP in eastern Uganda.

Study Objective: To determine the difference in the effectiveness of positive deviance and parent facilitator training strategies to malnutrition and caregiving among children and youth with cerebral palsy in the Iganga Mayuge and Bugweri districts.

Study setting: The study will be conducted within the districts of Iganga, Mayuge and Bugweri in eastern Uganda.

Study design: This will be a 2x2 factorial quasi-randomised controlled trial assessing the effects of the Positive deviance (PD) (Yes/No) and Parent facilitator training (PFT) (Yes/No) strategies within four experimental conditions: i) Both PD and PFT, ii) Only PD, iii)Only PFT, iv) Neither PD and nor PFT(controls).

Study population: The study population will include caregivers of malnourished children and youth aged 2-24 years old with a confirmed diagnosis of CP.

ELIGIBILITY:
Inclusion Criteria:

* Malnourished children and youth (<-2sd in any of height for age, weight for age and body mass index for age z-scores) with CP
* Caregivers of malnourished children and youth with CP

Exclusion Criteria:

* Caregivers registered in other nutrition interventions
* severely malnourished children that require life-saving nutrition management

Ages: 2 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 124 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2022-12-17 (Actual)

PRIMARY OUTCOMES:
Nutritional status | 3 months
  Mean weight gain

CONTACTS AND LOCATIONS:
Locations (1):
- Makerere University School of Public Health, Kampala, Uganda